CLINICAL TRIAL: NCT05989412
Title: Mobile Screening for Major Depressive Disorder in Adults From an Ethnically and Socioeconomically Diverse Population.
Acronym: MOOD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Inge MCM de Kok, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NL84280.078.23
Record Dates: First submitted 2023-05-09; First posted 2023-08-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: Randomized controlled trial; Major depressive disorder; Screening intervention; eHealth; Mental health
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will randomize 1786 eligible respondents across three arms, in a 2:1:1 fashion. The three arms comprise a control arm, a screening arm with limited participant referral for treatment (after three positive test scores on Patient Health questionnaire-9 (PHQ-9) or suicidal ideation), and a screening arm with standard referral for participants with moderate-severe symptoms of major depression (single positive test score on PHQ-9 questionnaire).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (No Intervention): a control arm where the investigators will only measure the quality of life using the EQ-5D questionnaire. This measurement will be performed at the same time as both screening arms.
- Standard referral (Experimental): a screening arm with standard participant referral for diagnosis at the general practitioner's office (after 1 positive test score on the PHQ-9 questionnaire or suicidal ideation).
  Interventions: Other: Patient health questionnaire-9 via the Your Research application
- Limited referral (Experimental): a screening arm with limited participant referral for diagnosis at the general practitioner's office (after three consecutive positive test scores on the PHQ-9 questionnaire or suicidal ideation).
  Interventions: Other: Patient health questionnaire-9 via the Your Research application

INTERVENTIONS:
Other: Patient health questionnaire-9 via the Your Research application — Both intervention arms will have 4-weekly screening with either lenient follow-up or screening with stricter follow-up for a time period of one year. Data will be collected via an app designed by Your Research which runs on Microsoft Azure server, as the primary of participants' response collection. A dedicated backup system will serve as a secondary data collection.
  Arms: Limited referral; Standard referral

SUMMARY:
Major depressive disorder (MDD) is a mental disorder leading to a variety of emotional and physical problems affecting almost 300 million people worldwide. Long-term treatments for MDD, including medication and therapy, imposes a significant financial burden on society. Mobile-based screening interventions might be a promising approach for effectively reducing MDD symptoms. The investigators hypothesize that the mobile-based screening strategy evaluated in this proposal will substantially reduce the burden of MDD over time, increase participants' quality of life, and decrease MDD-related disparities

DETAILED DESCRIPTION:
The MOOD trial is designed as a prospective, randomized controlled multi-arm trial with three parallel groups: an intervention group that will be screened 4-weekly for MDD for 12 months and receives a referral for MDD diagnosis and treatment after one positive test score on the PHQ-9, an intervention group who will be screened the same as the first group but receives a referral for MDD diagnosis and treatment after three consecutive positive test scores on the PHQ-9 and a control group who do not receive mobile-based screening for MDD. Randomization will be performed by the Your Research application as block randomization with a 2:1:1 allocation and stratification for age, gender and living area.

The intervention will be powered to demonstrate an effect on quality of life after 12 months with 80% power at a 5% significance threshold. It assumes that averted MDD will result in a 0.40 improvement in quality of life and that frequent screening will be effective in 40% of participants with MDD. Furthermore, the investigators conservatively assume a cumulative incidence of MDD during 12 months of 10%, based on a three times increased rate of unemployment in the intervention area and therefore three times increased risk of developing MDD. An additional adjustment for an assumed 40% spontaneously remission rate within 12 months was applied. With a correlation coefficient of 0.8, the design effect for using the baseline measurement becomes 0.36. Therefore, 714 people are required in control and combined intervention arms. Yielding a total sample size of 1,428 people (2:1:1 randomization). The intervention will be powered to demonstrate an effect on quality of life with 80% power at a 5% significance threshold. To compensate for the potential 20% differential loss of follow-up in both arms due to adverse events, the investigators aim to recruit an additional 179 participants for the control arm and 179 participants for the intervention arm (1:1 between both intervention groups). To reach the goal this study therefore need 1786 participants.

Participants will follow the individual screening procedure through the application platform Your Research. Participants will be invited to create a secured personal account, after which all participants can log in through a website on their computer/laptop or by installing the Your Research app on their tablet or mobile phone. There will be a variety of platforms provided for additional inquiries about the study process, including video calls, chat options, and phone calls.

Participants will be recruited through different online and offline strategies to encourage citizens' participation according to different cultural backgrounds. Offline recruitment includes in-person interactions with community members referred to be "key figures", posting flyers in GP offices and municipal buildings, video promotion, presentations, and by addressing people personally in public areas. Online recruitment postings will be made on websites, social media networks, and local radio stations.

Interested individuals can enroll by visiting the study website, or by initiating an application procedure through the Your Research app. If preferred, contacting the investigators through phone or email is also possible. Eligible participants will subsequently be provided with the patient information form (PIF) as well as an informed consent form. Participants who complete and return the signed consent form will be enrolled and randomized in the trial. The informed consent procedure is conducted digitally by using ValidSign. After randomization, participants will complete the baseline assessment.

Recruitment will be closely monitored to ensure that the sample size will be reached. If the sample size is attained, inclusion tactics will be discontinued. Furthermore, to ensure that questionnaire assessments are completed and that participants remain in the study, researchers will automatically send reminders via several contact channels based on the participants' preferences (email, push notifications, SMS). Participants will be compensated for their participation at the end of the study. Depending on the study arm and the number of completed questionnaires the participants can earn up to €50 in gift cards. Participants have the option to withdraw from the study at any moment during the trial. Recruitment will take place between January 2024 and December 2024.

Primary and secondary outcome measures for the MOOD study will be collected using mobile-based questionnaires. Data can be collected throughout the study and stored using encrypted digital files within password-protected folders with access limited to a restricted number of researchers. To protect confidentiality, participants will be granted a unique participant identification number upon registration. This number, as well as the associated personal information, is only available to the lead investigator and team members under their supervision. Contact information will be kept separate from any other research data gathered throughout the study. After the study is finished, all data will be safely archived for 15 years within Erasmus Medical Center. Once all outcome data has been collected, it will be exported to a statistics program. Members of the research team will examine and clean the data. All data will be kept and stored in accordance with the Personal Data Protection Act.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old Live in Rotterdam Zuid
* Have access to a smartphone or tablet.
* Give informed consent

Exclusion Criteria:

- Is currently treated by a psychologist or psychiatrist for depressive symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1786 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores after 12 months | 12 months
  Primary outcomes of the trial include participants' quality of life after 12 months as measured by the The 5-level EuroQuol-5D (EQ-5D-5L) between two intervention groups and the control group. EQ-5D-5L is being used as a 5-item self-report validated questionnaire for assessing health and health-related quality of life across five core dimensions (5D): mobility, self-care, daily activities, pain/discomfort, and anxiety/depression and has been widely used to measure the quality of life. Items are scored on zero-five levels of severity (5L) for each dimension. Higher scores represent decreased quality of life on that particular day with a minimum score of 5 and a maximum score of 25.

SECONDARY OUTCOMES:
Major depressive disorder symptoms | 12 months
  The investigators will also examine the occurrence and severity of symptoms as measured by the PHQ-9. If participants are not referred to their GP due to one or three consecutive positive test scores on PHQ-9 during the 12-month intervention period, PHQ-9 will be evaluated every four weeks for both intervention groups. Furthermore, population differences will be evaluated based on socio-demographic characteristics (including age, gender, ethnicity, education level, and employment status).
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression including 9 questions and a 4-scale-based answer option (Not at all, Several days, More than half the days, Nearly every day). Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively. Scores on the PHQ-9 range from 0 to 27. A higher score means a worse outcome

OTHER OUTCOMES:
Quality of life follow up | 24 months
  Other study parameters include participants' quality of life after 24 months as measured by the EQ-5D-5L between two intervention groups and the control group.
  EQ-5D-5L is being used as a 5-item self-report validated questionnaire for assessing health and health-related quality of life across five core dimensions (5D): mobility, self-care, daily activities, pain/discomfort, and anxiety/depression and has been widely used to measure the quality of life. Items are scored on zero-five levels of severity (5L) for each dimension. Higher scores represent decreased quality of life on that particular day with a minimum score of 5 and a maximum score of 25.

CONTACTS AND LOCATIONS:
Overall Officials: Inge de Kok, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data of participants that did not grant permission to reuse their data for future research will have to be removed. Furthermore, further pseudonymisation and/or aggregation of the pseudonymised dataset would be required to secure the privacy of the participants and avoid indirect identification.
  The accessibility of the collected data could be important for potential follow-up research of this project and/or similar national/international projects that would like to perform analyses on our data because not much is known yet on the implementation of screening for MDD.
Supporting Information: Study Protocol
Time Frame: The data will be published within 10 months and will be available from then on.
Access Criteria: Open source publication

REFERENCES:
- [Background] Abdoli N, Salari N, Darvishi N, Jafarpour S, Solaymani M, Mohammadi M, Shohaimi S. The global prevalence of major depressive disorder (MDD) among the elderly: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2022 Jan;132:1067-1073. doi: 10.1016/j.neubiorev.2021.10.041. Epub 2021 Nov 4. PMID 34742925
- [Background] Almeida OP. Prevention of depression in older age. Maturitas. 2014 Oct;79(2):136-41. doi: 10.1016/j.maturitas.2014.03.005. Epub 2014 Mar 22. PMID 24713453
- [Background] Gotlib IH, Goodman SH, Humphreys KL. Studying the Intergenerational Transmission of Risk for Depression: Current Status and Future Directions. Curr Dir Psychol Sci. 2020 Apr 1;29(2):174-179. doi: 10.1177/0963721420901590. Epub 2020 Feb 24. PMID 33758474
- [Background] Hall CA, Reynolds-Iii CF. Late-life depression in the primary care setting: challenges, collaborative care, and prevention. Maturitas. 2014 Oct;79(2):147-52. doi: 10.1016/j.maturitas.2014.05.026. Epub 2014 Jun 7. PMID 24996484
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Kalibatseva Z, Leong FT. Depression among Asian Americans: Review and Recommendations. Depress Res Treat. 2011;2011:320902. doi: 10.1155/2011/320902. Epub 2011 Sep 27. PMID 21961060
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Liu Q, He H, Yang J, Feng X, Zhao F, Lyu J. Changes in the global burden of depression from 1990 to 2017: Findings from the Global Burden of Disease study. J Psychiatr Res. 2020 Jul;126:134-140. doi: 10.1016/j.jpsychires.2019.08.002. Epub 2019 Aug 10. PMID 31439359
- [Background] O'Connor EA, Whitlock EP, Beil TL, Gaynes BN. Screening for depression in adult patients in primary care settings: a systematic evidence review. Ann Intern Med. 2009 Dec 1;151(11):793-803. doi: 10.7326/0003-4819-151-11-200912010-00007. PMID 19949145
- [Background] Park LT, Zarate CA Jr. Depression in the Primary Care Setting. N Engl J Med. 2019 Feb 7;380(6):559-568. doi: 10.1056/NEJMcp1712493. PMID 30726688
- [Background] Posternak MA, Miller I. Untreated short-term course of major depression: a meta-analysis of outcomes from studies using wait-list control groups. J Affect Disord. 2001 Oct;66(2-3):139-46. doi: 10.1016/s0165-0327(00)00304-9. PMID 11578666
- [Background] Rohde P, Lewinsohn PM, Klein DN, Seeley JR, Gau JM. Key Characteristics of Major Depressive Disorder Occurring in Childhood, Adolescence, Emerging Adulthood, Adulthood. Clin Psychol Sci. 2013 Jan;1(1):10.1177/2167702612457599. doi: 10.1177/2167702612457599. PMID 24273703
- [Background] Siu AL; US Preventive Services Task Force (USPSTF); Bibbins-Domingo K, Grossman DC, Baumann LC, Davidson KW, Ebell M, Garcia FA, Gillman M, Herzstein J, Kemper AR, Krist AH, Kurth AE, Owens DK, Phillips WR, Phipps MG, Pignone MP. Screening for Depression in Adults: US Preventive Services Task Force Recommendation Statement. JAMA. 2016 Jan 26;315(4):380-7. doi: 10.1001/jama.2015.18392. PMID 26813211
- [Background] Sobocki P, Jonsson B, Angst J, Rehnberg C. Cost of depression in Europe. J Ment Health Policy Econ. 2006 Jun;9(2):87-98. PMID 17007486
- [Background] Steensma C, Loukine L, Orpana H, McRae L, Vachon J, Mo F, Boileau-Falardeau M, Reid C, Choi BC. Describing the population health burden of depression: health-adjusted life expectancy by depression status in Canada. Health Promot Chronic Dis Prev Can. 2016 Oct;36(10):205-213. doi: 10.24095/hpcdp.36.10.01. PMID 27768557
- [Background] Whiteford HA, Harris MG, McKeon G, Baxter A, Pennell C, Barendregt JJ, Wang J. Estimating remission from untreated major depression: a systematic review and meta-analysis. Psychol Med. 2013 Aug;43(8):1569-85. doi: 10.1017/S0033291712001717. Epub 2012 Aug 10. PMID 22883473
- [Background] Yildiz B, Schuring M, Knoef MG, Burdorf A. Chronic diseases and multimorbidity among unemployed and employed persons in the Netherlands: a register-based cross-sectional study. BMJ Open. 2020 Jul 2;10(7):e035037. doi: 10.1136/bmjopen-2019-035037. PMID 32616488
- [Derived] Zandbergen MME, Jansen EEL, Jabbarian LJ, de Koning HJ, de Kok IMCM. A mobile-based randomized controlled trial on the feasibility and effectiveness of screening for major depressive disorder: study protocol. BMC Psychol. 2024 Dec 18;12(1):742. doi: 10.1186/s40359-024-02230-6. PMID 39695914